CLINICAL TRIAL: NCT03248180
Title: Impact of Guided Antipsychotic Dose Reduction in Patients With Psychosis Under Remitted States: a Randomized Control Trial and Prospective Follow-up Study
Brief Title: Guided Dose Reduction of Antipsychotic in Patients With Psychosis in Remitted States
Acronym: GDR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201703002MIND
Record Dates: First submitted 2017-08-06; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Psychosis; Remission
Keywords: antipsychotic; guided dose reduction; maintenance treatment; remitted psychosis; relapse
MeSH Terms: conditions — Psychotic Disorders; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma for determining concentration of antipsychotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Guided dose reduction (GDR): Patients in the GDR group will be advised to reduce < 25% of their current dose of antipsychotic agents estimated on a weekly base and follow-up every 4 weeks for at least 12 weeks.
- Maintenance treatment group (MTG): Patients in the MTG will be advised to stay on their current dose of antipsychotics throughout the observational period, follow-up every 12 weeks.

SUMMARY:
A 2-year prospective observational study comparing a group of patients in remitted states of psychosis undergoing guided antipsychotic dose reduction to a similar group of patients under maintenance antipsychotic treatment with the main outcome of interest that if the rates of relapse of psychosis between these two groups will be different.

DETAILED DESCRIPTION:
Early intervention at the beginning of schizophrenia and related psychotic disorders can get better treatment response. Once symptoms subsided, the majority of patients wish to discontinue medications, yet currently the mainstream opinions still recommend maintenance antipsychotic therapy because non-adherence to medication is the most significant risk factor to predict a relapse. However, recent longitudinal studies assessing patients in community for a longer term found that their functioning is not necessarily poorer despite not regularly treated with antipsychotics. Also there are studies suggesting a lower percentage of dopamine occupancy by antipsychotic is acceptable in stable patients with psychosis. To elucidate such discrepancies, a hypothetical compromised approach "guided dose reduction, but not aiming at discontinuation"is proposed. In this study, we will recruit outpatients with schizophrenia related psychotic disorders under remitted states, randomize into guided dose reduction group (GDR, n = 80) and maintenance treatment group (MTG), including those who willing to have dose reduction but assigned to maintenance group (MTG1, n = 40) and those who willing to continue medication serving as naturalistic observation group (MTG2, n = 40), and follow up for at least 2 years. The main outcomes of interests are differences in relapse rates, personal social performance, quality of life, drug-related adverse reactions, medication satisfaction, and neurocognitive function between groups.We will also have patients to keep logs of medication status, blood tests for therapeutic drug monitoring, biochemistry, and potential biomarkers, as well as take into account demographic variables such as age, gender, education, employment status, and supportive system, and clinical variables such as age of onset, duration of illness, history of psychiatric admission, the highest and the lowest doses of antipsychotics during previous treatment, the number of different antipsychotics having being tried before, if a history of impending relapse during tapering down dose of antipsychotics, and concomitant psychotropic agents, to test whether these variables are related to outcomes during follow-up. Hopefully we can identify a satisfactory and balanced solution between improving patient's psychosocial and neurocognitive outcomes and prevention of relapse by redefining the role of antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of schizophrenia, schizophreniform disorder, psychosis NOS, based on the DSM-5 criteria
2. With a Positive and Negative Syndrome Scale (PANSS), score < 3 in all 3 positive symptoms (P1: delusion, P2: conceptual disorganization, P3: hallucination) and 2 general symptoms (G9: unusual thought, G5: mannerism and posturing) for at least 3 months
3. With a PANSS score < 4 in all 3 negative symptoms (N1: blunted affect, N4: social withdrawal, N6: lack of spontaneity/flow in conversation) for at least 3 months
4. Currently receiving antipsychotic treatment at a fixed dose for at least 3 months, including long-acting injectable antipsychotic
5. A second antipsychotic agent only used for a low-dose, as needed adjuvant purpose
6. No revised use of benzodiazepines, antidepressants, anticholinergics, or other concomitant medications during past 3 months -

Exclusion Criteria:

1. A score of 5 or more on any of the 30 PANSS rating items at screening
2. Admission to acute psychiatric unit during past 6 months
3. A change in dose of current antipsychotic medication in recent 3 months
4. Concomitant use of mood stabilizers, such as lithium, valproic acid or other anti-epileptic drugs
5. Mental retardation known as IQ below 70 prior to the diagnosis of schizophrenia
6. A history of pervasive mental disorder or bipolar disorder
7. A medical condition with significant cognitive sequelae
8. A history of substance dependence during past 6 months
9. Currently in pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Outpatients received follow-up at or referred to the study hospital
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse of psychosis defined by worsening of scores in Positive and Negative Syndrome Scale (PANSS) | up to 2 years
  Patients will be measured with a Positive and Negative Syndrome Scale (PANSS) every 4 weeks for 3 times (during 12 weeks) if conducting dose reduction or every 12 weeks if staying on the same dose to observe if any worsening of symptoms. Patient has a PANSS score > 4 in any item of those 3 positive symptoms (P1: delusion, P2: conceptual disorganization, P3: hallucination) and 2 general symptoms (G9: unusual thought, G5:mannerism and posturing) during observational period for more than 1 week will be recognized as having a relapse of psychosis.

SECONDARY OUTCOMES:
Personal Social Performance (PSP) scores | up to 2 years
  Patients will be rated by their attending psychiatrists with PSP scale to evaluate their functioning in 4 aspects of life, including socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviors as to give a summary score at baseline and annually
quality of life (Euro-5D VAS) | up to 2 years
  Patients report their quality of life using a 20-cm visual analogue at baseline and annually.
severity of extrapyramidal symptoms | up to 2 years
  Patient's severity of extrapyramidal symptoms will be rated by their psychiatrists using Simpson-Angus Scale, the Abnormal Involuntary Movement Scale, and the Barnes Akathisia Rating Scale at each visit.
medication satisfaction questionnaire (MSQ) | up to 2 years
  Patients will be asked to fill a self-rated 7-point Likert scale for medication satisfaction at baseline and annually.
neurocognitive functioning | up to 2 years
  Patients will be assessed with the module for schizophrenia of the Cambridge Neuropsychological Test Automatic Battery (Cantab) at baseline and at the exit of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Chung Liu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan